CLINICAL TRIAL: NCT01872507
Title: The Effect of Breathing Biofeedback Training to Influence the Function of the Cardiac Autonomic Nervous System at Rest and in Activity in Children With Cerebral Palsy.
Brief Title: BioFeedBack Breathing Training Influence Cardiac Autonomic Nervous System in Children With Cerebral-Palsy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, BERGER ITAI, Director Neuro-Cognitive Center Pediatric Wing, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMO-0374-12
Record Dates: First submitted 2013-05-01; First posted 2013-06-07 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Cerebral Palsy; Autonomic Nerveus System
Keywords: cerebral palsy; autonomic nerveus system; heart rate variability
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- biofeedback training (Active Comparator): usual treatment+12 treatment of biofeedback training
  Interventions: Other: Biofeedback training
- control (No Intervention): usual treatment

INTERVENTIONS:
Other: Biofeedback training — usual treatment +12 biofeedback training
  Arms: biofeedback training

SUMMARY:
The effect of breathing biofeedback training to influence the function of the cardiac autonomic nervous system at rest and in activity in children with cerebral palsy.

Cerebral palsy children suffer from a non-progressive damage of the brain. It is the most common injury that causes physical handicapped in childhood. There are a few researches that investigated the autonomic function in cerebral palsy children. Those researches found hyperactivity of the sympathetic autonomic system, including high resting heart rate compare to their typically developed pears. The recommended treatment for cerebral palsy is activity, muscle strengthening and mobility. The impairment in the autonomic system influences the everyday function and has correlation with secondary morbidity.

As far as we know there are no researches who investigated the following issues.

In this study we would like to:

1. Describe the autonomic cardiac function, Breathing function, motor function and the correlation between them in children with cerebral palsy.
2. Compare the autonomic cardiac function at rest in aerobic test and in diaphragmatic breathing.
3. Test the influence of breathing training on Heart rate variability parameters at rest, in aerobic test right after the breathing training program and one month after, in children with cerebral palsy

DETAILED DESCRIPTION:
Participants:

60 children with cerebral palsy age 6-11 who can walk and understand simple instructions.

Main outcome measures:

Heart rate variability using Polar watch and transmitter RS810CX.

Secondary outcome measures:

1. Lung functioning using Sensormedics Vmax 29 spirometry:Forced Vital Capacity, Forced Expiratory Volume in one,Tidal Volume.
2. Biofeedback
3. Sub maximal aerobic test on treadmill-Modified Naughton Protocol with Polar watch and transmitter.
4. Gross Motor Function Classification System
5. Gross Motor Function Measure
6. Functional Mobility Scale
7. Children Assessment of Participation and Enjoyment
8. Autonomic function questionnaire

ELIGIBILITY:
Inclusion Criteria:

* children with cerebral palsy
* age 6-11 years
* able to walk
* both gender

Exclusion Criteria:

* heart or lung known disease
* can not follow simple commends

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of Heart rate variability meaures at one and two months | Change from Baseline at one and two months

SECONDARY OUTCOMES:
Change from Baseline of Forced Vital Capacity, Forced Expiratory Volume in one, Tidal Volume, | Change from Baseline at one and two month
Change from Baseline Sub maximal aerobic test on treadmill-Modified Naughton Protocol with Polar watch and transmitter. | Change from baseline at one and two month later
Change from baseline breathing rate, by biofeedback | Change from baseline at one and two month later

OTHER OUTCOMES:
Change from baseline Gross Motor Function Measure | Change from baseline at one and two month later
Change from baseline Children Assessment of Participation and Enjoyment | Change from baseline at one and two month later
Change from baseline Autonomic function questionnaire | Change from baseline at one and two month later

CONTACTS AND LOCATIONS:
Overall Officials: Itai Berger, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Zamuner AR, Cunha AB, da Silva E, Negri AP, Tudella E, Moreno MA. The influence of motor impairment on autonomic heart rate modulation among children with cerebral palsy. Res Dev Disabil. 2011 Jan-Feb;32(1):217-21. doi: 10.1016/j.ridd.2010.09.020. Epub 2010 Oct 16. PMID 20956067
- [Background] Sutarto AP, Wahab M, Zin NM. Heart Rate Variability (HRV),biofeedback; A new training approch for aperator's performance enhancement. JIEM, 2010, 3;176-198.
- [Background] Ferreira MC, Pastore C, Imada R, Guare R, Leite M, Poyares D, Santos MT. Autonomic nervous system in individuals with cerebral palsy: a controlled study. J Oral Pathol Med. 2011 Aug;40(7):576-81. doi: 10.1111/j.1600-0714.2011.01008.x. Epub 2011 Feb 16. PMID 21323740
- [Background] Lehrer PM, Vaschillo E, Vaschillo B. Resonant frequency biofeedback training to increase cardiac variability: rationale and manual for training. Appl Psychophysiol Biofeedback. 2000 Sep;25(3):177-91. doi: 10.1023/a:1009554825745. PMID 10999236